CLINICAL TRIAL: NCT04041609
Title: A Phase II, Randomized, Blinded, Sham Procedure-Controlled, Parallel-Group Trial to Evaluate the Efficacy, Safety and Tolerability of LYR-210 in Adult Subjects With Chronic Sinusitis (LANTERN Study)
Brief Title: LYR-210 Depot (LYR-210) for Adult Subjects With Chronic Sinusitis (LANTERN Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lyra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYR-210-2018-002; 2018-004621-89 (EudraCT Number)
Record Dates: First submitted 2019-07-12; First posted 2019-08-01 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-05

CONDITIONS: Chronic Sinusitis; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LYR-210 (Low Dose) (Experimental): In-office bilateral placement of the LYR-210 drug depot (mometasone furoate low dose) in the middle meatus
  Interventions: Drug: LYR-210
- LYR-210 (High Dose) (Experimental): In-office bilateral placement of the LYR-210 drug depot (mometasone furoate high dose) in the middle meatus
  Interventions: Drug: LYR-210
- Sham Procedure (Sham Comparator): In-office bilateral sham procedure
  Interventions: Other: Sham comparator

INTERVENTIONS:
Drug: LYR-210 — A single administration of LYR-210 depot
  Arms: LYR-210 (High Dose); LYR-210 (Low Dose)
Other: Sham comparator — Sham comparator
  Arms: Sham Procedure

SUMMARY:
This is a Phase II, Randomized, Blinded, Sham Procedure-Controlled, Parallel-Group Trial to Evaluate the Efficacy, Safety and Tolerability of LYR-210 in Adult Subjects with Chronic Sinusitis.

DETAILED DESCRIPTION:
LYR-210 is a drug depot, which contains the anti-inflammatory medication mometasone furoate (MF) pre-loaded in a single use applicator. LYR-210 is intended to be placed bilaterally into the sino-nasal passages by an otolaryngologist. Once in place, each LYR-210 drug depot is designed to gradually deliver sustained topical doses of MF to the inflamed mucosal sinus tissue over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CS.
* Two trials of medical treatments for CS in the past.
* Minimum CS symptom score.
* Ability to tolerate topical anesthesia.
* Has been informed of the nature of the study and has provided written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site.
* Agrees to comply with all study requirements.

Exclusion Criteria:

* Have undergone previous sinus surgery.
* Pregnant or breast feeding.
* Known history of hypersensitivity or intolerance to corticosteroids.
* History or clinical evidence or suspicion of invasive fungal sinusitis, allergic fungal rhinosinusitis, or atrophic rhinitis.
* Known history of hypothalamic pituitary adrenal axial dysfunction or having a morning serum cortisol level at screening outside of the normal range.
* Had dental procedure/implant on maxillary dentition within 4 weeks of the Screening visit.
* Past or present functional vision in only one eye.
* Has cataracts
* Past, present, or planned organ transplant or chemotherapy with immunosuppression.
* Currently participating in an investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Australia (4):
  - Royal Brisbane and Woman's Hospital, Brisbane
  - Monash Health, Clayton
  - The ENT Centre, Hornsby
  - Westmead Hospital, Westmead
- University Hospital for Otorhinolaryngology, Medical University of Graz, Vienna, Austria
- Czechia (4):
  - Fakultní nemocnice Plzeň, Pilsen, Czech Republic
  - Fakultni Nemocnice Hradec Kralove Klinika otorinolaryngologie a chirurgie hlavy a krku, Hradec Králové, Prague
  - Fakultni Nemocnice Brno OR, Brno
  - St Anne's Faculty Hospital, Brno
- New Zealand (7):
  - Southern Clinical Trials Waitemata, Auckland
  - Southern Clinical Trials Ltd, Christchurch
  - Clinical Trials New Zealand, Hamilton
  - Middlemore Clinical Trials, Papatoetoe
  - P3 Research Tauranga, Tauranga
  - P3 Research Wellington, Wellington
  - Wellington Hospital, Wellington
- Poland (6):
  - Provita Sp. z o.o. Centrum Medyczne Angelius Provita, Katowice
  - Centrum Medyczne All-Med, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne PROMED, Krakow
  - Centrum Zdrowia MDM, Warsaw
  - Vistamed Sp. z o.o., Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided
All Individual Participant Data (IPD) that underlie results in a publication may be available to other researchers.

REFERENCES:
- [Background] Cervin A, Rimmer J, Wrobel A, Abelak Y, Brayton L, Kuang Y. Long-acting implantable corticosteroid matrix for chronic rhinosinusitis: Results of LANTERN Phase 2 randomized controlled study. Int Forum Allergy Rhinol. 2022 Feb;12(2):147-159. doi: 10.1002/alr.22883. Epub 2021 Sep 17. PMID 34534410

RESULTS

PARTICIPANT FLOW:
Groups:
- LYR-210 (Low Dose): In-office bilateral placement of the LYR-210 drug depot (mometasone furoate 2500 µg) in the middle meatus
  LYR-210: A single administration of LYR-210 depot
- LYR-210 (High Dose): In-office bilateral placement of the LYR-210 drug depot (mometasone furoate 7500 µg) in the middle meatus
  LYR-210: A single administration of LYR-210 depot
Period: Overall Study
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Started | 24 | 23 | 24
Completed | 17 | 15 | 17
Not Completed | 7 | 8 | 7

BASELINE CHARACTERISTICS:
Population: The primary analysis set for efficacy is the Intent-to-treat (ITT) set which includes all randomized subjects who received the study treatment and had a post-Day 1 assessment available.
Groups:
- Total: Total of all reporting groups
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure | Total
Number analyzed (Participants) | 23 | 21 | 23 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (12.72) | 46.9 (12.72) | 41.3 (14.68) | 43.4 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 12 | 32
  Male | 11 | 13 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 21 | 23 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 21 | 22 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 1 | 1 | 3
  Australia | 4 | 2 | 2 | 8
  Europe | 18 | 18 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFBL) in Chronic Sinusitis Symptom Scores at Week 4
Description: Participants score their CS symptoms on a 4-point scale as follows: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom present but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping). The scores are summed and averaged over the proceeding 7 days; higher scores indicate higher severity of symptoms of CS.
Time Frame: Week 4
Population: ITT analysis set: all randomized subjects who receive the study treatment or have a treatment attempt on Day 1 and have post-Day 1 assessments available
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 23 | 21 | 23
score on a scale | -2.24 (0.637) | -2.65 (0.651) | -2.28 (0.611)

2. Secondary Outcome: Change From Baseline in the 22-item Sino-nasal Outcome Test (SNOT-22) Total Score at Week 24
Description: Participants score the severity of their symptoms and social/emotional consequences of CS on a 6-point scale: 0 = no problem, 1 = very mild problem, 2 = mild or slight problem, 3 = moderate problem, 4 = severe problem, 5 = problem as bad as it can be. The scores are summed in the range of 0-110; higher scores indicate higher severity of symptoms or social/emotional consequences of CS.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 23 | 21 | 23
score on a scale | -30.0 (5.32) | -40.7 (5.76) | -21.7 (5.10)

3. Secondary Outcome: CFBL in Chronic Sinusitis Symptom Scores at Week 24
Description: as for outcome 1
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 23 | 21 | 23
score on a scale | -3.36 (0.668) | -4.32 (0.682) | -2.68 (0.640)

4. Secondary Outcome: Participants With Improved Bilateral Zinreich Score at Week 24
Description: Each sinus is assigned a score based on the percentage of opacification as follows: 0 = 0%, 1 = 1% to 25%, 2 = 26% to 50%, 3 = 51% to 75%, 4 = 76 % to 99%, 5 = 100% or completely occluded. Each sinus pair has a bilateral score in the range of 0 to 10. Higher scores indicate higher severity of sinus opacification. Responder is defined as a participant with at least a 1-point decrease in the imaging score at Week 24 compared with baseline.
Time Frame: Week 24
Population: The outcome measure is based on the Intent-to-treat (ITT) set which includes all randomized subjects who received the study treatment and had a post-Day 1 imaging assessment which could be analyzed by the imaging core lab.
Measure: Count of Participants; unit: Participants
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 19 | 19 | 18
Participants | 13 | 14 | 10

5. Secondary Outcome: The Number of Participants With Treatment-related Adverse Events for up to 24 Weeks
Description: To evaluate the safety and tolerability of LYR-210
Time Frame: 24 weeks
Population: The safety analysis population contains all subjects who were randomized and either received the study treatment (Sham or either dose of LYR-210) or had a treatment attempt on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 24 | 23 | 23
Participants | 11 | 5 | 5

6. Secondary Outcome: Plasma Drug Concentrations of MF at Week 4
Description: To evaluate the pharmacokinetics of LYR-210
Time Frame: 4 Weeks
Population: Participants who had evaluable plasma concentration at week 4.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 20 | 16 | 0
pg/mL | 13.6110 (5.21710) | 45.3500 (11.40783) |

7. Secondary Outcome: Plasma Drug Concentrations of MF at Week 12
Description: To evaluate the pharmacokinetics of LYR-210
Time Frame: 12 weeks
Population: Participants who had evaluable plasma concentration at week 12.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
Number analyzed (Participants) | 16 | 14 | 0
pg/mL | 21.6500 (7.77869) | 30.9143 (12.04657) |

ADVERSE EVENTS:
Time Frame: 1 year
Description: AEs are collected from the time of informed consent until week 48/EOS visit. The safety analysis population contains all subjects who were randomized and either received the study treatment (Sham or either dose of LYR-210) or had a treatment attempt on Day 1.
Arm/Group | LYR-210 (Low Dose) | LYR-210 (High Dose) | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 15/24 | 13/23 | 12/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYR-210 (Low Dose) (N=24) | LYR-210 (High Dose) (N=23) | Sham Procedure (N=23)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LYR-210 (Low Dose) (N=24) | LYR-210 (High Dose) (N=23) | Sham Procedure (N=23)
Facial Pain (General disorders) | 1 | 2 | 0
Chronic Sinusitis (Infections and infestations) | 4 | 4 | 7
Rhinitis (Infections and infestations) | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04041609/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT04041609/SAP_001.pdf